CLINICAL TRIAL: NCT03041727
Title: Physiotherapist Approach to Shoulder's Diseases, Differences Between Fascial Manipulation and Standard Exercise
Brief Title: Physiotherapist Approach to Shoulder's Diseases, Differences Between Fascial Manipulation and Standard Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Bolognini di Seriate Bergamo (Other)
Responsible Party: Principal Investigator, silvia Bellotti, Physiotherapist, Azienda Ospedaliera Bolognini di Seriate Bergamo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOBolognini 1
Record Dates: First submitted 2017-01-27; First posted 2017-02-03 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Shoulder Pain; Manual Therapy
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study are evaluated in parallel against a control group.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be a statistic techinician, with any knowledge about the group composition and the rehabilitative intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Group (Active Comparator): The subjects will be treated with a standard protocol of stretching and strengthening exercises , we require them to do the exercises by themselves during five weeks, one a day.
  To make sure that they will do the protocol, we'll give them a diary to sign the daily section.
  Interventions: Other: Standard exercises protocol
- Intervention group (Experimental): The subjects will be treated with the same protocol of the Standard Group, but in two section, they will receive a Fascial Manipulation approach.
  Interventions: Other: Fascial Manipulation

INTERVENTIONS:
Other: Fascial Manipulation — Fascial Manipulation is a manual therapy that focused on deep muscular fascial.
  Arms: Intervention group
Other: Standard exercises protocol — Stretching and strengthening exercises
  Arms: Standard Group

SUMMARY:
The study purpose is to compare the effects of Fascial Manipulation added to standard exercises protocol versus the simple exercises protocol.

DETAILED DESCRIPTION:
The shoulder degenerative diseases are recurring in hospital employees. The early approach, as we see in literature, has high probability to reduce the pain and the disfunction in the long term.

In particular stretching and strengthening exercises are the standard protocol applied.

The Fascial Manipulation is a manual therapy that works on the connective tissue, by increasing mobility and reducing pain.

We have added the Fascial Manipulation to prove if it make a faster recovery and a pain reduction in the short and the middle term.

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain and acute and relapse in six months
* positive results in two orthopedic testes

Exclusion Criteria:

* Degenerative diseases and neurological diseases
* Rheumatological Diseases and cancer
* fracture of the humerus, scapula and collarbone
* documented injury of rotator cuff.
* cortisones therapy in action

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain | Before and after the first treatment. A week after the enrollment.
  VNS scale in the Apley 'Scratch Test

SECONDARY OUTCOMES:
shoulder' function | Before and after the first treatment. A week after the enrollment.
  Constant Morley Scale
shoulder' function | Before and after the fifth treatment, after five weeks. This will be the last treatment
  Constant Morley Scale
shoulder' function | A month later the last treatment, as follow up
  Constant Morley Scale
Range of Movement of the shoulder | Before and after the first treatment. A week after the enrollment.
  Bubble Inclinometer used in the flexion, abduction and external rotation movement
Range of Movement of the shoulder | Before and after the fifth treatment, after five weeks.This will be the last treatment
  Bubble Inclinometer used in the flexion, abduction and external rotation movement
Range of Movement of the shoulder | A month later the last treatment, as follow up
  Bubble Inclinometer used in the flexion, abduction and external rotation movement
The shoulder's muscular strength | Before and after the first treatment. A week after the enrollment.
  dynamometer survey in flexion and abduction movement
The shoulder's muscular strength | Before and after the fifth treatment, after five weeks. This will be the last treatment
  dynamometer survey in flexion and abduction movement
The shoulder's muscular strength | A month later the last treatment, as follow up
  dynamometer survey in flexion and abduction movement

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Busato, first level, Study Director — Azienda Ospedaliera Bolognini di Seriate Bergamo
Locations (1):
- AO Bolognini, Seriate, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No